CLINICAL TRIAL: NCT06067763
Title: Enhancing Effectiveness of a Dissonance-Based Obesity Prevention Program: Randomized Controlled Trial
Brief Title: Project Health: Enhancing Effectiveness of an Obesity Prevention Program
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: Stanford University (Other); Drexel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HD093598
Record Dates: First submitted 2023-09-22; First posted 2023-10-05 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Overweight and Obesity; Eating Disorders
Keywords: obesity; overweight; eating disorders; prevention; adolescent; dissonance
MeSH Terms: conditions — Overweight; Obesity; Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be masked to participant condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Female Group, Food Response Training (Experimental): Participants in this arm will be assigned to receive Project Health in female-only groups and will complete the food-focused response and attention training intervention.
  Interventions: Behavioral: Project Health; Behavioral: Response and Attention Training
- Male Group, Food Response Training (Experimental): Participants in this arm will be assigned to receive Project Health in male-only groups and will complete the food-focused response and attention training intervention.
  Interventions: Behavioral: Project Health; Behavioral: Response and Attention Training
- Educational Video control (Active Comparator): Participants in this arm will be assigned to watch a four-part documentary "The Weight of the Nation" from their home.
  Interventions: Other: The Weight of the Nation

INTERVENTIONS:
Behavioral: Project Health — A brief dissonance-based obesity prevention program delivered in six one-hour weekly sessions.
  Arms: Female Group, Food Response Training; Male Group, Food Response Training
Behavioral: Response and Attention Training — Individualized, computerized response and attention training consisting of five separate tasks designed to increase inhibitory control to reduce overeating.
  Arms: Female Group, Food Response Training; Male Group, Food Response Training
Other: The Weight of the Nation — This 2012 documentary discusses the facts and myths about obesity and the impacts of obesity on individuals and the health care system in the United States.
  Arms: Educational Video control

SUMMARY:
This 2-site effectiveness trial will test whether a brief dissonance-based obesity prevention program delivered in single sex groups combined with food response and attention training will produce significantly larger weight gain prevention effects than an educational video control condition. An effectiveness trial is important to test whether this program reduces risk for unhealthy weight gain when delivered by real world clinicians under ecologically valid conditions, which is an important step toward broad implementation. A secondary aim focuses on eating disorder symptom prevention effects. A sample of 17-20 year olds with weight concerns (N = 120) will be randomized to single sex Project Health groups with food response and attention training or an educational video control condition. Participants will complete assessments at baseline, posttest, and 6- and 12-month follow ups.

DETAILED DESCRIPTION:
In the previous Project Health trial, the investigators found Project Health is most effective when implemented in single sex groups paired with food specific response and attention training. This project will evaluate the effectiveness of this version of the Project Health intervention compared to a video control condition and is an important step toward dissemination. A brief effective obesity prevention program that can be easily, inexpensively, and broadly implemented to late adolescents at risk for excess weight gain, as has been the case with another dissonance-based prevention program, could markedly reduce the prevalence of obesity and associated morbidity and mortality. The program may also have an important secondary benefit of preventing the onset of future eating symptoms and disorders. The study has 2 aims: (1) Test the hypothesis that Project Health implemented in single-sex groups and paired with food response inhibition and attention training produces significantly larger weight gain and overweight/obesity onset prevention effects than an educational video control condition (primary outcome). (2) Test the hypothesis that Project Health implemented in single-sex groups and paired with food response inhibition and attention training produces significantly larger eating disorder symptom prevention effects than an educational video control condition (secondary outcome).

ELIGIBILITY:
Inclusion Criteria:

* Current at least moderate weight concerns (defined as a response of 4 or above on an 8 point scale ranging from none (0) to extreme (8))
* Self-reported room for improvement in diet and exercise habits (response of yes to "Do you believe there is room for improvement in your diet and exercise habits?" in the pre-screening questionnaire)
* BMI greater than or equal to 20 and less than or equal to 30
* Age between 17 and 20 years old

Exclusion Criteria:

* Current diagnosis of anorexia nervosa, bulimia nervosa or binge eating disorder
* Previous participation in a Project Health study

Ages: 17 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 238 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Body Fat | baseline, posttest (approximately 8 weeks after baseline), 6-month follow-up (approximately 34 weeks after baseline), 12-month follow-up (approximately 60 weeks after baseline)
  Change in percentage of body fat as measured by air displacement plethysmography (ADP) via the Bod Pod.

SECONDARY OUTCOMES:
Eating Disorder Symptoms | baseline, posttest (approximately 8 weeks later), 6-month follow-up (approximately 34 weeks after baseline), 12-month follow-up (approximately 60 weeks after baseline)
  The Eating Disorder Diagnostic Interview, a brief semi-structured interview will assess eating disorder symptoms. It provides diagnoses for anorexia nervosa, bulimia nervosa, and binge eating disorder. It also provides a continuous measure of overall eating disorder symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Oregon Research Institute, Springfield, Oregon

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share all study data via the NICHD Data and Specimen Hub (DASH), which is the centralized resource for researchers to store and access data from NICHD-funded research studies to use for secondary research. All data, with the exception of video recordings of the participants in treatment (which cannot be effectively de-identified), will be provided.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After all follow-up assessments are completed and the main project papers are published, a dataset stripped of identifiers prior to release will be made available without cost to researchers and analysts.